CLINICAL TRIAL: NCT03315325
Title: Age-dependent Changes in the Responsiveness of Hypothalamic Pituitary Gonadal Axis to Kisspeptin-10 Administration in Men
Brief Title: Age-dependent Changes in the Responsiveness of Hypothalamic Pituitary Gonadal Axis in Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Quaid-e-Azam University (Other)
Responsible Party: Principal Investigator, Ghulam Nabi, Doctoral Researcher, Quaid-e-Azam University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Quaid-i-Azam University
Record Dates: First submitted 2017-09-30; First posted 2017-10-20 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Sterility, Reproductive
Keywords: Aging
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Healthy men, 15 in number were selected. These individuals were classified on the basis of their ages in three groups: adult, middle age and advanced aged. Each group comprised of five participants.
Masking Description: There was no masking. Every individual was told about injecting the kisspeptin, however, they were not informed at the time when kisspeptin was injected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adult men (Experimental): The average age was 25.80±0.37 years and intervention human kisspeptin-10 was administered in single iv bolus dose (1 µg/kg BW). Serial blood samples were collected for 30 min pre and 120 min post-kisspeptin injection periods at 30 min interval.
  Interventions: Biological: Human kisspeptin-10 (metastin 45-54)
- Middle age men (Experimental): The average age was 47.00±0.77 years and intervention human kisspeptin-10 was administered in single iv bolus dose (1 µg/kg BW). Serial blood samples were collected for 30 min pre and 120 min post-kisspeptin injection periods at 30 min interval.
  Interventions: Biological: Human kisspeptin-10 (metastin 45-54)
- Advance age men (Experimental): The average age was 73.20±0.91 years and intervention human kisspeptin-10 was administered in single iv bolus dose (1 µg/kg BW). Serial blood samples were collected for 30 min pre and 120 min post-kisspeptin injection periods at 30 min interval.
  Interventions: Biological: Human kisspeptin-10 (metastin 45-54)

INTERVENTIONS:
Biological: Human kisspeptin-10 (metastin 45-54) — Kisspeptin-10 (metastin 45-54, Calbiochem, Darmstadt, Germany) is a potent HPG-axis stimulator and control reproduction.

SUMMARY:
The present study was designed to assess the responsiveness of the hypothalamic pituitary gonadal axis to kisspeptin administration with increasing age in men.

DETAILED DESCRIPTION:
Little is known about the involvement of kisspeptin signalling in the causation of senescence-basal modulation of the GnRH-LH unit in any model and particularly in advance age men. The present study was therefore designed to assess the response of hypothalamic pituitary gonadal axis to kisspeptin administration with increasing age in healthy men. Sequential blood samples (2 ml) were obtained for 30 minutes pre and 120 minutes post-kisspeptin injection periods at 30 min intervals (-30, 0, 30, 60, 90, 120). Kisspeptin-10 was administered (1 µg/kg BW) as an intravenous bolus, immediately after collecting 0 min sample to assess the response of GnRH neurons to kisspeptin-10 with increasing age in men by determining plasma levels of LH and testosterone.

ELIGIBILITY:
Inclusion Criteria:

• Age

Exclusion Criteria:

* Hepatic and renal complications
* Epilepsy
* Pneumonia
* Asthma
* Orchitis
* Hernia
* Cryptorchidism
* Cardiovascular diseases
* Reproductive disorders
* Mental retardation

Ages: 25 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-08-08 (Actual); Primary Completion 2014-08-10 (Actual); Study Completion 2015-03-05 (Actual)

PRIMARY OUTCOMES:
To investigate the basal function of KISS1R on GnRH neurons through serum LH and testosterone during aging in men | Two blood samples at 30 minutes interval before kisspeptin injection were obtained from all the groups to determine basal levels for LH and testosterone.
Changes in the sensitivity of KISS1R by determining the responsiveness of GnRH neuron to kisspeptin administration after 30 minutes during aging in men through measuring plasma luteinizing hormone and testosterone concentrations | One blood sample from all individuals were obtained after 30 minutes of post kisspeptin injection for measuring a change in LH and testosterone.
Changes in the sensitivity of KISS1R by determining the responsiveness of GnRH neuron to kisspeptin administration after 60 minutes during aging in men through measuring plasma luteinizing hormone and testosterone concentrations | One blood sample from all individuals were obtained after 60 minutes of post kisspeptin injection for measuring a change in LH and testosterone.
Changes in the sensitivity of KISS1R by determining the responsiveness of GnRH neuron to kisspeptin administration after 90 minutes during aging in men through measuring plasma luteinizing hormone and testosterone concentrations | One blood sample from all individuals were obtained after 90 minutes of post kisspeptin injection for measuring a change in LH and testosterone.
Changes in the sensitivity of KISS1R by determining the responsiveness of GnRH neuron to kisspeptin administration after 120 minutes during aging in men through measuring plasma luteinizing hormone and testosterone concentrations | One blood sample from all individuals were obtained after 120 minutes of post kisspeptin injection for measuring a change in LH and testosterone.

CONTACTS AND LOCATIONS:
Overall Officials: Shahab, Study Chair — Quaid-i-Azam University
Locations (1):
- Quaid-i-Azam University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
After publishing will be available to all researchers. Additional data will be provided by the corresponding author on request.

REFERENCES:
- [Result] Chan YM, Butler JP, Pinnell NE, Pralong FP, Crowley WF Jr, Ren C, Chan KK, Seminara SB. Kisspeptin resets the hypothalamic GnRH clock in men. J Clin Endocrinol Metab. 2011 Jun;96(6):E908-15. doi: 10.1210/jc.2010-3046. Epub 2011 Apr 6. PMID 21470997
- [Result] Dhillo WS, Chaudhri OB, Patterson M, Thompson EL, Murphy KG, Badman MK, McGowan BM, Amber V, Patel S, Ghatei MA, Bloom SR. Kisspeptin-54 stimulates the hypothalamic-pituitary gonadal axis in human males. J Clin Endocrinol Metab. 2005 Dec;90(12):6609-15. doi: 10.1210/jc.2005-1468. Epub 2005 Sep 20. PMID 16174713
- [Result] George JT, Veldhuis JD, Roseweir AK, Newton CL, Faccenda E, Millar RP, Anderson RA. Kisspeptin-10 is a potent stimulator of LH and increases pulse frequency in men. J Clin Endocrinol Metab. 2011 Aug;96(8):E1228-36. doi: 10.1210/jc.2011-0089. Epub 2011 Jun 1. PMID 21632807
- [Result] Jayasena CN, Nijher GM, Comninos AN, Abbara A, Januszewki A, Vaal ML, Sriskandarajah L, Murphy KG, Farzad Z, Ghatei MA, Bloom SR, Dhillo WS. The effects of kisspeptin-10 on reproductive hormone release show sexual dimorphism in humans. J Clin Endocrinol Metab. 2011 Dec;96(12):E1963-72. doi: 10.1210/jc.2011-1408. Epub 2011 Oct 5. PMID 21976724